CLINICAL TRIAL: NCT06206343
Title: Comparison of the Effectiveness of Telerehabilitation With Transcutaneous Electrical Nerve Stimulation on Pain and Functionality in Individuals With Chronic Neck Pain: Randomized Controlled Trial
Brief Title: Telerehabilitation With Transcutaneous Electrical Nerve Stimulation Chronic Neck Pain:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, MUSA ÇANKAYA, Lecturer Doctor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MCANKAYA
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Chronic Neck Pain; Telerehabilitation; Transcutaneous Electrical Nerve Stimulation; Pain
Keywords: Neck Pains; Tele-rehabilitation; Transcutaneous Electric Stimulation,; Chronic Pain
MeSH Terms: conditions — Pain; Neck Pain; Chronic Pain | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Posttest and control grouped randomized controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: 45
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TENS application treatment program (Experimental): Conventional TENS will be performed for 3 weeks and 15 sessions. In this application, two electrodes will be placed on each side of the spinous processes of the patient's cervical region.
  Two of them will be placed right and left, just below the skull, where the scalp ends, and the other two will follow them, about 5 cm away.
  Care will be taken not to place the electrodes directly on your spine.
  Interventions: Other: TENS application, Tele-rehabilitation treatment program
- Tele-rehabilitation application treatment program: (Experimental): Patients who accept the treatment will be evaluated before treatment. The treatment program will be done online for 3 weeks, 3 times a week. In the first session, neck anatomy and things to be considered in neck pain will be explained to the patient. In the following sessions, neck exercises will be performed with the participation of the patients.
  Neck exercises: 1.Head rotation movements 2.Chin tuck 3.Neck isometric exercises 4.Shoulder shrug 5.Scapula approach 6.Isometric strengthening 7.Exercises against gravity 8.Stretching exercises etc. will be done.
  Interventions: Other: TENS application, Tele-rehabilitation treatment program
- Control group (No Intervention): Control group patients will not receive any treatment. The first evaluation was done.
  After 3 weeks, the second evaluation will be done again.

INTERVENTIONS:
Other: TENS application, Tele-rehabilitation treatment program — Exercise training
  Other Names: Exercise training:
  Arms: TENS application treatment program; Tele-rehabilitation application treatment program:

SUMMARY:
Nonspecific chronic neck pain (NCNP) is defined as non-specific neck pain lasting more than three months. It is a very common disease that causes a great obstacle in the daily life activities of individuals in the society. Many conservative treatment methods are used in the treatment of this disease. Among these treatment methods, Transcutaneous Electrical Nerve Stimulation (TENS) is the most widely used modality due to its low cost and many advantages. There are 4 types of TENS: Conventional, Low frequency (Acupuncture), Short intensity, Combined or Burst TENS. Conventional TENS is generally used in the treatment of chronic pain.

Tele-rehabilitation is defined as the delivery of rehabilitation services via online telecommunication technologies. Tele-rehabilitation overcomes many problems such as long distance, traffic, transportation difficulties, high cost, high demand in the public health system, etc. and its popularity is increasing with the developments in technology and telecommunications. The risks and difficulties of accessing physical treatment during the COVID-19 pandemic have demonstrated the necessity of Tele-rehabilitation. Therefore, Tele-rehabilitation is widely used in physiotherapy as well as in many other fields.

Although TENS application is widely used in the treatment of nonspecific chronic neck pain in physiotherapy clinics, there are few studies on Tele-rehabilitation, there are no studies comparing their effectiveness compared to each other in this field. In our research, it is planned to investigate and compare the effectiveness of TENS, which is an easily applied electrotherapy method, and Tele-Rehabilitation, an online rehabilitation tool. In this study, the staff of Nezahat Keleşoğlu Faculty of Health Sciences and Seydişehir Vocational School of Health Services and patients with neck pain who come to the physiotherapy unit of Meram Medical Faculty Hospital will be included in the study. As a result of the power analysis, (48) patients are planned to be included.

Patients will be divided into three as Tele-rehabilitation group and TENS group and Control group. Patients will be evaluated before and after treatment and training.

DETAILED DESCRIPTION:
Nonspecific chronic neck pain (NCNP) is a highly prevalent disorder that causes a major impediment to individuals' activities of daily life. It is largely influenced by psychosocial factors. This disease is defined as pain in the lateral and posterior neck without pathologic symptoms lasting more than 12 weeks(1). The number of common cases of neck pain worldwide is estimated to be 288.7 million, and the worldwide prevalence of this disorder (16.7% to 75.1%) has been reported(2,3).The incidence is higher in women than men (4).

The mechanisms underlying the progression of NKBA are not clear, but it is thought to be related to impaired proprioception of the neck muscles, which play a decisive role in cervical joint position and motor control of the head (5). Spinal manipulation, acupuncture, massage therapy, exercise, traction, soft cervical collar, electrotherapy, yoga and Tele-rehabilitation are the modalities used in the treatment of this disease (6-14).

One of the most basic applications among these is Transcutaneous electrical nerve stimulation (TENS). TENS is one of the modalities commonly used to relieve pain in the musculoskeletal system(4). TENS is the most preferred electroanalgesia method because it is easy to apply, has few side effects, is relatively safe, non-invasive, low-cost and can be easily applied by patients at home. TENS provides pain relief through the physiologic pathways of low-voltage electric current produced by electrodes adhered to the skin. Gate control theory, hyperstimulation analgesia and endorphin metabolism are used to reduce pain (15,16,17).

Models used in Tens therapy:

* Conventional TENS: It is applied in the form of pulses with high frequency (50-100 Hz) and low current passage time. It creates a needling and tingling sensation in the painful area. The effect of conventional TENS starts within 30 minutes and disappears 2 hours after treatment.
* Low frequency (Acupuncture) TENS: produces visible muscle contraction and has a low frequency (1-5Hz) and high current transit time. Acupuncture TENS increases the release of endorphins by affecting small diameter C fibers and produces an analgesic effect.
* Short intensity TENS: It is short-intensity and intense, with a frequency of more than 100 Hz and produces pulses of wide width and intensity up to the patient's highest tolerance. In this model, all sensory and motor fibers are affected. Analgesia effect starts in 1-15 minutes and disappears in a short time after stimulation.
* Combined or Burst TENS: This model is a combination of high (50-100 Hz) and low (1-10 Hz) frequency currents. Muscle contraction is visible and the analgesic effect starts later and lasts longer.

The most commonly used models in TENS treatment are conventional TENS and acupuncture TENS (18,19).Conventional TENS will be applied to the patients in our study.

Tele-rehabilitation is defined as the delivery of rehabilitation services through telecommunication technologies such as websites, smartphone applications, online video conferencing systems (20). Tele-rehabilitation is a suitable platform to provide services in the field of physiotherapy as it is used in many fields.Today, tele-rehabilitation is increasing in popularity with advances in technology and telecommunications, overcoming some of the potential barriers to access to health care such as distance, traffic, transportation difficulties, high cost, high demand in the public health system (long waiting lists), lack of insurance coverage for private health care (21,22).

The risks and difficulties of accessing physical treatment during the COVID-19 pandemic have revealed the necessity of tele-rehabilitation(23). Tele-rehabilitation has been used in many physiotherapy fields such as pediatrics, pneumology, musculoskeletal pain and neurology, but few studies have examined its effect on neck pain(24).

Despite the widespread use of TENS in the treatment of nonspecific chronic neck pain in physiotherapy clinics, there have been few studies on Tele-rehabilitation, and there are no studies comparing their effectiveness compared to each other in this field. In our research, it is planned to investigate the ethics of TENS, an easy-to-apply electrotherapy method, and Tele-Rehabilitation, an online rehabilitation tool. Therefore, the aim of the present study was to investigate the comparative effectiveness of Tele-rehabilitation training or TENS therapy on pain, functionality and quality of life in patients with NKBA.

Patients who come to Meram Medical Faculty Physical Therapy Unit will be included in this study. In addition, Necmettin Erbakan University Nezahat Keleoğlu Faculty of Health Sciences, Kamil Akkanat Faculty of Health Sciences students and employees who have neck pain for more than 3 months and do not have disc herniation etc. will be included.

ELIGIBILITY:
Inclusion Criteria:

* Being between 18-55 years old
* People with non-specific neck pain, defined as pain not attributed to a cause
* Neck pain that has persisted for at least three months and recurs more than 1 time,
* Agreeing to participate in the study,
* To be able to read and write Turkish
* Have a computer, tablet or smartphone and an active internet connection,
* Having at least 2 points of pain according to the Visual Analog Scale at rest, and having a score of 10 and above according to the Neck Disability Index,
* Being able to use a computer, tablet and the internet at a level to participate in video conferencing or having a relative who can help in this regard (10,23,25,27)

Exclusion Criteria:

Spinal surgery history

* Traumatic cervical injuries
* Serious comorbidities (neurological, neuromuscular, cardiological, psychiatric)
* Cervical region fractures
* Tumoral conditions
* Having vision and hearing problems
* Cognitive influences
* People with skin allergies
* Scleroderma, vasculitis or neuropathic pathologies
* People with pacemakers
* Pregnant women (10,23,25)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Bournemouth neck pain questionnaire | valuation will be made before and after treatment. The evaluation is expected to take 10 minutes in total.
  This questionnaire consists of 7 questions in total. Developed in 2002 in the UK. It includes questions about pain, disability and psychosocial issues (33). Each question is scored between 0 and 10. The highest score is 70 and the closer the score is to 70, the higher the patient's level of disability. The content of the questionnaire consists of variables such as pain severity, the effect of pain on activities of daily living and social life, anxiety-depression level, kinesiophobia and coping with pain. The Turkish version of the questionnaire was conducted by Telci et al. (34).
Neck Disability Index (NDI) | valuation will be made before and after treatment. The evaluation is expected to take 10 minutes in total
  The NDI was designed by Vernon and Mion to assess how neck pain affects functionality related to activities of daily living (42). In a 3-year prospective study conducted for the prediction of long-term health problems after neck injury, only the NDI was associated with true significance. Furthermore, in cross-cultural studies conducted in French, Swedish (albeit modified), Portuguese and Dutch, the NDI has proven to be a valid and reliable tool for measuring disability (43). The Turkish validity and reliability of the scale was conducted by Aslan et al. (2009) (44,45).
Copenhagen Neck Functional Disability Scale (CNFDS) | valuation will be made before and after treatment. The evaluation is expected to take 10 minutes in total
  It is a scale completed by the patient. It was developed in 1998 by Jordan. The questionnaire consisting of 15 questions evaluates the severity of pain, activities of daily living, social and recreational activities, and the future status of neck pain.Questions 1, 2, and 3 in this questionnaire evaluate attention; questions 4 and 5 evaluate proprioceptive sensation; questions 6, 7, and 9 evaluate the perception of neck shape and size; and question 8 evaluates neglect.The total score in this questionnaire varies between 0-30, and an increase in score indicates an increase in the level of disability (35, 36).
World Health Organization Quality of Life Module (WHOQOL-BREF) | valuation will be made before and after treatment. The evaluation is expected to take 10 minutes in total
  WHOQOL, a general purpose quality of life profile scale, has two versions, long and short. The health-related quality of life scale was developed by WHO and its validity and reliability was performed by Eser et al. The scale has two versions, long (WHOQOL-100) and short (WHOQOL-27). The scale measures physical, mental, social and environmental well-being and consists of 26 questions (37). The scale can be applied to non-elderly adults. The scale has also been applied to healthcare professionals. Since each domain independently expresses the quality of life in its own domain, domain scores are calculated between 4-20. The higher the score, the better the quality of life (38).

CONTACTS AND LOCATIONS:
Overall Officials: Musa Çankaya, Pt.PhD., Principal Investigator — Necmettin Erbakan University; Sami Küçükşen, Prof.Dr., Principal Investigator — Necmetin Erbakan University, MeramFacultyofMedicine; PARİYA POURİYAMANESH, Int.Pt, Principal Investigator — Necmettin Erbakan University
Locations (1):
- Musa Çankaya, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Cankaya M, PourIYamanesh P, Kucuksen S. Investigation of the effectiveness of interactive telerehabilitation and transcutaneous electrical nerve stimulation on pain, functionality, disability and quality of life in patients with nonspecific chronic neck pain: a randomised controlled trial. Expert Rev Med Devices. 2025 Mar;22(3):243-252. doi: 10.1080/17434440.2025.2471444. Epub 2025 Feb 26. PMID 39988923